CLINICAL TRIAL: NCT00951808
Title: Preventing Acute Chest Syndrome by Transfusion Feasibility Study( PROACTIVE Feasibility Study)
Brief Title: Preventing Acute Chest Syndrome by Transfusion Feasibility Study
Acronym: PROACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 668; U10HL083721 (NIH)
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Results first posted 2013-04-05 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Sickle Cell Disease
Keywords: Anemia, Sickle Cell; Acute Chest Syndrome; Secretory phospholipase A2(sPLA2)
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome | interventions — Blood Transfusion; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Blood Transfusion Trial Cohort (Active Comparator): Twenty participants will receive a blood transfusion while in the hospital.
  Interventions: Biological: Single blood transfusion
- Standard Care Trial Cohort (Active Comparator): Twenty participants will not receive a blood transfusion and will receive standard care.
  Interventions: Behavioral: Standard care
- Standard Care Observational Cohort (Active Comparator): Approximately 300 participants who are ineligible for or decline the blood transfusion part of the study will participate in the observational portion of the study and receive standard care.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Biological: Single blood transfusion — Participants will receive a single transfusion of 7-13cc/kg packed red blood cells (RBCs) while in the hospital.
  Other Names: transfusion
  Arms: Blood Transfusion Trial Cohort
Behavioral: Standard care — Participants will receive standard care for ACS while in the hospital.
  Other Names: standard of care
  Arms: Standard Care Observational Cohort; Standard Care Trial Cohort

SUMMARY:
Acute chest syndrome (ACS) is similar to severe pneumonia and is a common cause of hospitalizations for people with sickle cell disease (SCD). Blood transfusions are one treatment option for ACS. High levels of an enzyme called secretory phospholipase A2 (sPLA2) may be present in people before they develop ACS. This study will determine how well sPLA2 levels can predict the onset of ACS and whether identifying high sPLA2 levels allows enough time to prevent ACS with blood transfusions. Results from this study will help to determine the feasibility of conducting a larger study that would further examine the use of sPLA2 levels and blood transfusions to prevent ACS in people with SCD.

DETAILED DESCRIPTION:
SCD is an inherited blood disorder, and symptoms include anemia, infections, organ damage, and intense episodes of pain, which are called "sickle cell crises." ACS, characterized by fever, respiratory distress, and lung tissue damage, is the second most common cause of hospitalization and the leading cause of death among people with SCD. Most people with SCD will experience at least one episode of ACS, and repeated episodes can result in progressive lung disease. ACS can appear suddenly and often requires immediate hospitalization and treatment, which can include blood transfusions. People with elevated blood levels of sPLA2 may be at risk for developing ACS, and this enzyme is often detectable before the onset of ACS symptoms. The purpose of this study is to examine the use of sPLA2 as a predictor of ACS and to determine whether subsequent blood transfusions can be administered early enough to prevent the onset of ACS in people with SCD who are at risk for ACS. Study researchers will also assess the feasibility of conducting a larger study that would further examine the effectiveness of using sPLA2 levels and blood transfusions to prevent ACS.

This study will involve two parts. In the first part of the study, participants with SCD who are admitted to the hospital with an acute sickle cell pain event will be randomly assigned to receive either a single blood transfusion or standard care for ACS and no blood transfusion. All participants will be closely monitored while in the hospital for the development of ACS, and study researchers will review participants' medical records. All participants will undergo daily blood collections, which will include testing for sPLA2 levels, and at least two chest x-rays. Twenty-eight days after hospital discharge, all participants will attend a follow-up study visit for blood collection, again to determine sPLA2 levels.

In the second part of the study, participants who are not eligible or who do not choose to participate in the first part of the study will be enrolled into an observational group. These participants will receive standard care for ACS, but will not receive a blood transfusion. They will undergo daily blood collection during their hospital stay and at least one chest x-ray. While participants are in the hospital and 28 days after discharge, study researchers will review participants' medical records.

ELIGIBILITY:
Inclusion Criteria for the Observational and Trial Cohorts:

* Hemoglobin diagnosis of SS (two copies of the hemoglobin S gene), SC (one copy of the hemoglobin S gene and one copy of the hemoglobin C gene), or S-β thalassemia (β+ or β0)
* No clinically apparent ACS
* No prior participation in either part of the study

Inclusion Criteria for the Trial Cohort, in addition to the above criteria:

* sPLA2 level greater than 100 ng/mL within the same 24-hour window that coincides with fever and chest radiograph negative for new pulmonary infiltrate within the last 12 hours of the 24-hour window
* Fever greater than 38.0º C within the same 24-hour window that coincides with elevated sPLA2 level (greater than 100 ng/mL) and chest radiograph negative for new pulmonary infiltrate within the last 12 hours of the 24-hour window
* Chest radiograph negative for new pulmonary infiltrate within the last 12 hours of the 24-hour window of an abnormal sPLA2 level and fever
* Hemoglobin levels equal or less than 10 g/dL at time of study entry
* Informed consent of parent(s) or legal guardian; informed consent or assent of participant as applicable

Exclusion Criteria for Observational and Trial Cohorts:

* Existing diagnosis of a new pulmonary infiltrate diagnosed by chest radiography (pleural effusion not obscuring lung parenchyma will not exclude the person from the study)
* Any coexisting medical condition for which the physician feels that a transfusion may be needed within 24 hours (e.g., severe anemia, stroke)
* Red Blood Cell (RBC) transfusion in the 60 days before study entry
* Unwillingness to sign consent form, or if a minor, unwillingness of parent/guardian to sign consent form
* Treatment with any investigational drug or device in the 30 days before study entry (hydroxyurea is allowable)
* History of alloimmunization that would prevent the participant from receiving blood within 8 hours of eligibility for study entry or history of a life-threatening transfusion reaction
* Objection to transfusion for religious or other reasons from either the participant or guardian
* History of treatment with systemic steroids within 1 week of study entry (inhaled steroids are acceptable)
* Pregnant

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja McKinlay, PhD, Principal Investigator — Carelon Research; Margaret C. Bell, MPH, MS, Study Director — Carelon Research
Locations (24):
- United States (24):
  - Children's Hospital and Research Center, Oakland, California
  - A.I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Illinois Sickle Cell Center, Chicago, Illinois
  - Kosair Children's Hospital, Louisville, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Interfaith Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Virginia Commonwealth University Health Systems, Richmond, Virginia

REFERENCES:
- [Result] Miller ST, Kim HY, Weiner D, Wager CG, Gallagher D, Styles L, Dampier CD; Investigators of the Sickle Cell Disease Clinical Research Network (SCDCRN). Inpatient management of sickle cell pain: a 'snapshot' of current practice. Am J Hematol. 2012 Mar;87(3):333-6. doi: 10.1002/ajh.22265. Epub 2012 Jan 9. PMID 22231150
- [Result] Styles L, Wager CG, Labotka RJ, Smith-Whitley K, Thompson AA, Lane PA, McMahon LE, Miller R, Roseff SD, Iyer RV, Hsu LL, Castro OL, Ataga KI, Onyekwere O, Okam M, Bellevue R, Miller ST; Sickle Cell Disease Clinical Research Network (SCDCRN). Refining the value of secretory phospholipase A2 as a predictor of acute chest syndrome in sickle cell disease: results of a feasibility study (PROACTIVE). Br J Haematol. 2012 Jun;157(5):627-36. doi: 10.1111/j.1365-2141.2012.09105.x. Epub 2012 Mar 30. PMID 22463614
- [Derived] Miller ST, Kim HY, Weiner DL, Wager CG, Gallagher D, Styles LA, Dampier CD, Roseff SD; Investigators of the Sickle Cell Disease Clinical Research Network (SCDCRN). Red blood cell alloimmunization in sickle cell disease: prevalence in 2010. Transfusion. 2013 Apr;53(4):704-9. doi: 10.1111/j.1537-2995.2012.03796.x. Epub 2012 Jul 13. PMID 22804353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the period June 2009 - June 2010, 237 subjects from 25 sites were enrolled in the feasibility study. Of 237 enrolled, only 10 were randomized (six subjects in the Standard Care Arm and four subjects in the Transfusion Arm). The randomization trial has been terminated due to the lack of enrollment.
Groups:
- Blood Transfusion Trial Cohort: Subjects received a transfusion within 6 hours of randomization.
- Standard Care Trial Cohort: Subjects received standard care (regular care for acute chest syndrome (ACS)) without a clinically indicated transfusion.
- Standard Care Observational Cohort: Subjects who are ineligible for or who decline the blood transfusion part of the study participated in the observational portion of the study and received standard care (regular care for acute chest syndrome (ACS)).
Period: Overall Study
Arm/Group | Blood Transfusion Trial Cohort | Standard Care Trial Cohort | Standard Care Observational Cohort
Started | 4 | 6 | 227
Completed | 4 | 6 | 223 (Four subjects withdrew from the study.)
Not Completed | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The randomization trial has been terminated due to the lack of enrollment. Therefore, the results were not reported by Arm and the total number of subjects (237) enrolled in the feasibility study was used.
Groups:
- All Participants: 237 subjects enrolled in the feasibility study.
Arm/Group | All Participants
Number analyzed (Participants) | 237
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 122
  Between 18 and 65 years | 114
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119
  Male | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 230
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3
  Black or African American | 230
  More than one race | 1
  Other | 3
Maximum secretory phospholipase A2 (sPLA2) value [Number; unit: participants] — Maximum secretory phospholipase A2 (sPLA2) value measured prior to acute chest syndrome (ACS) or discharge
  participants
    >0 - 25 ng/ml | 106
    >25 - 50 ng/ml | 34
    >50 - 100 ng/ml | 22
    >100 - 200 ng/ml | 13
    >200 - 800 ng/ml | 28
    Not applicable | 34

OUTCOME MEASURES:

1. Primary Outcome: Acute Chest Syndrome
Description: First occurence of positive infiltrate on chest x-ray
Time Frame: Chest x-rays (CXR) were ordered for trial eligibility, as a result of clinical indications, or at discharge or 72 hours if no prior CXR.
Population: Of 237 enrolled subjects, 27 subjects who received a transfusion and 7 subjects who had insufficient sPLA2 measurements were excluded. Therefore, two hundred and three (203) subjects were included in the analysis. Results were not reported by Arm due to the lack of enrollment.
Measure: Number; unit: participants
Groups:
- Adults: Age >= 18
- Children: Age < 18
- Overall: Both adults and children
Arm/Group | Adults | Children | Overall
Number analyzed (Participants) | 96 | 107 | 203
participants
  Yes | 11 | 11 | 22
  No | 85 | 96 | 181
Statistical Analysis 1: Comparison: Adults vs Children vs Overall; The optimal threshold level (TL), determined via receiver operating characteristic (ROC) curve analysis, maximizes the difference between the true positive rate (TPR) and the false positive rate (FPR). Since there is no corresponding analytic standard deviation (SD) for this value, we computed a robust SD based upon the interquartile range (IQR)/1.35 from a bootstrap sample of optimal TLs; Test type: Superiority or Other; optimal threshold level of sPLA2 = 48, 95% CI 2-sided [38 to 58], Standard Deviation 5 — The optimal threshold level (TL) was determined to be the same for all analysis groups

ADVERSE EVENTS:
Description: According to the protocol, adverse events (AEs) were only reportable for subjects who received a trial-indicated transfusion (blood transfusion trial cohort). Due to the early termination and low enrollment for the randomization trial, we are not reporting results for this cohort. Therefore, there are no AEs to report.
Arm/Group | Blood Transfusion Trial Cohort
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The feasibility study has been completed, but the randomization trial has been terminated early due to the lack of enrollment. Therefore, the results were reported with the subjects who completed the feasibility study and were not reported by Arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes